CLINICAL TRIAL: NCT06367712
Title: The Effect of Using Letrozole Alone Protocol Versus Using Letrozole and HCG Protocol on Induction of Ovulation in Polycystic Ovarian Syndrome Patients: A Prospective Cohort Study
Brief Title: Letrozole Alone Protocol Versus Using Letrozole and HCG Protocol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ahmed Kassab
Record Dates: First submitted 2024-04-09; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: letrozole only (Active Comparator): About 66 Patients took Letrozole drug only for induction of ovulation at the time of suspected ovulation maturity.
  Interventions: Drug: Letrozole tablets
- Group B: letrozole + HCG (Active Comparator): About 66 Patients took Letrozole drug in addition to HCG for induction of ovulation at the time of suspected ovulation maturity.
  Interventions: Drug: Letrozole tablets

INTERVENTIONS:
Drug: Letrozole tablets — To determine if the usage of All interventions are effective for simple induction of ovulation in polycystic ovarian syndrome in infertile couples.
  Other Names: HCG

SUMMARY:
Letrozole is a chemical compound, CGS 20267 which is a third-generation, nonsteroidal aromatase inhibitor.

Letrozole blocks estrogen synthesis by directly affecting the hypothalamic-pituitary-ovarian axis, subsequently, increases gonadotropins which increase pregnancy rates. Possible positive outcomes of aromatase inhibitors over selective estrogen-receptor modulators include a more physiologic hormonal stimulation of the endometrium which increases receptivity, a lower multiple-pregnancy through single follicle growth, a lesser side-effect especially vasomotor and mood symptoms, and more prompt clearance from blood, hence, reducing the probabilities of periconceptional exposure

DETAILED DESCRIPTION:
The first pilot study for the clinical use of letrozole for ovarian induction in polycystic ovary syndrome (PCOS) patients was done in 2000.

In large randomized study, letrozole was superior to clomiphene as a treatment for anovulatory infertility in women with the polycystic ovary syndrome. Letrozole was also associated with higher live-birth and ovulation rates.

Ovulation induction with letrozole is associated with an ovulation rate of 70%-84% and a pregnancy rate of 20%-27% per cycle.

While in another study which Compare the Effect of Letrozole Alone with Letrozole Plus N-Acetylcysteine on Pregnancy Rate in Patients with Polycystic Ovarian Syndrome, the pregnancy rate was 7.5% in letrozole alone group .

Human chorionic gonadotropin (HCG) hormone will replace the naturally surging luteinizing hormone at mid-cycle, subsequently, will lead to full maturation of oocytes resulting in ovulation. Additionally, HCG will also enhance the endometrial quality by stimulating the corpus luteum. HCG is a hormone that is produced mainly by the placental syncytiotrophoblasts cells, it is also produced by other organs in minute amounts (Liver, colon and pituitary gland). HCG main function is maintaining pregnancy through stimulating the corpus luteum to produce progesterone.

This hormone is the cornerstone drug for inducing final maturation of follicles during a diversity of infertility treatment protocols.

In order to diagnose Polycystic ovarian syndrome two out of three Rotterdam criteria should be present. These criteria are: chronic anovulation, clinical and/or biochemical evidence of hyperandrogenism, and polycystic ovaries by ultrasound .

incidence of PCOS from 6% to 21% when the ESHRE/ASRM 2003 criteria were applied. Infertility (clinical definition) is currently defined as 1 year of unwanted non-conception with unprotected intercourse in the fertile phase of the menstrual cycles

ELIGIBILITY:
Inclusion Criteria:

* Infertile women with PCOS
* Normal hysterosalpingography
* Normal semen analysis according to WHO parameters are major prerequisites

Exclusion Criteria:

* Infertile women with causes other than PCOS,
* Ages <18 or >35 years
* women taken confounding medications like other infertility drugs
* Insulin sensitizers or hormones
* Abnormal hysterosalpingography
* Subnormal semen analysis

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Pregnancy test | 2 weeks after ovulation
  The participants required to make pregnancy test after taking the drugs of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher Teaching Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided